CLINICAL TRIAL: NCT06916858
Title: Prevalence of OSA and Diagnostic Accuracy of Type 3 Home Sleep Test in Difficult-to-treat Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0722/66
Record Dates: First submitted 2024-02-07; First posted 2025-04-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: OSA
Keywords: asthma; OSA; HSAT; home sleep test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Masking Description: mask the result of home sleep test and Polysonography
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- difficult to treat asthma (Other): difficult to treat asthma run HST and PSG
  Interventions: Device: home sleep test

INTERVENTIONS:
Device: home sleep test — Apnealink air
  Other Names: polysonography

SUMMARY:
cross sectional cohort study enroll Patients diagnosed with difficult-to-treat asthma, aged over 18 years, and experiencing persistent symptoms as assessed by the Asthma Control Test (ACT) underwent type 1 in-laboratory polysomnography and type 3 HSAT within 1 month apart

ELIGIBILITY:
Inclusion Criteria:

* difficult-to-treat asthma .
* Patients aged 18 years or older

Exclusion Criteria:

* Patients or volunteers unable to undergo type 1 and type 3 sleep studies,
* Patients with symptoms compatible with other sleep disorders,
* Patients with a history of or current stroke or transient ischemic attack and Other chronic respiratory diseases.
* Patients diagnosed with obstructive sleep apnea

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of OSA in patients with difficult-to-treat asthma | up to 4 months
  prevalence of OSA in patients with difficult-to-treat asthma

SECONDARY OUTCOMES:
assess the accuracy of type 3 home sleep apnea test (HSAT) | up to 1 months
  number of participant who have same diagnosed OSA with type 3 HSAT compare to type 1 sleep test
  * AHI
  * ODI

CONTACTS AND LOCATIONS:
Locations (1):
- Tidarat Somreusean, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided